CLINICAL TRIAL: NCT06079996
Title: Effects of Caffeinated Gum on a Batting and Pitching Performance of Female Softball Players: a Crossover Trial
Brief Title: Caffeinated Gum Softball Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chih-Hui Chiu (Other)
Responsible Party: Sponsor-Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 112-2
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Caffeine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine gum (Experimental): The gum containing 200 mg of caffeine (CAF) were chewed for 10 minutes before test
  Interventions: Other: CAFFEINE GUM
- placebo (Placebo Comparator): The gum without caffeine (PLA) were chewed for 10 minutes before test
  Interventions: Other: CAFFEINE GUM

INTERVENTIONS:
Other: CAFFEINE GUM — Observing the effect of chewing gum on the performance of female softball players.

SUMMARY:
The purpose of this study was to investigate the effects of caffeinated chewing gum on female softball pitching and hitting performance. 24 trained female softball players (10 pitchers and 14 fielders) were divided into a caffeine chewing gum trial (CAF) or a placebo trial (PLA) in a single-blind, randomized, crossover experimental design. Two pieces of gum containing 100 mg of caffeine (CAF) or without caffeine (PLA) were chewed for 10 minutes and then spit out, followed by a 15-minute warm-up. The physical tests included grip strength and countermovement jump. The softball-specific tests included pitching (fast ball speed) or hitting (exit speed). The two trials were separated by seven days.

DETAILED DESCRIPTION:
This study utilized a randomized, crossover, single-blind experimental design. At least two familiarization tests were conducted one week before the formal trial to ensure each participant was familiar with the experimental procedures. Before the first formal trial, participants were randomly assigned to either the caffeinated chewing gum trial (CAF) with 200 mg of caffeine or the placebo trial (PLA) without caffeine, seven days apart (Figure 1). The primary outcome was the pitching and hitting performance, and the secondary outcomes were hand grip strength and height of countermovement jump.

ELIGIBILITY:
Inclusion Criteria:

* 1. adult female; 2. at least six years of professional softball training and familiarity with all softball skills; 3. caffeine intake of less than 80 mg daily.

Exclusion Criteria:

* 1. not professionally trained; 2. having a medical condition for which exercise is not recommended, such as hypertension, hyperlipidemia, or heart disease; 3. having any musculoskeletal injuries within the last six months or not being able to complete a full trial; 4. having a history of caffeine allergy.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only professional female softball players
Enrollment: 24 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
pitching performance | 15 min after intervention
  Throw 10 fastballs
batting performance | 15 min after intervention
  Hit 15 balls

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-05-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT06079996/Prot_000.pdf